CLINICAL TRIAL: NCT06539416
Title: Leveraging Mixed Reality in MitraClip Implantation: a Preliminary Case Series Toward a Pilot Study
Brief Title: Mixed Reality in MitraClip Implantation: Preliminary Case Series
Acronym: MIMIC
Status: Recruiting | Type: Observational
Sponsor: Nemocnice AGEL Trinec-Podlesi a.s. (Other)
Responsible Party: Principal Investigator, Ing. Jan Hečko, Lead Biomedical Engineer, Nemocnice AGEL Trinec-Podlesi a.s.
Other Study IDs: INT2021011
Record Dates: First submitted 2024-07-25; First posted 2024-08-06 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-08

CONDITIONS: Mitral Regurgitation
Keywords: MitraClip,; MixedReality; Hololens; DICOM; Rendering; Support
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mixed Reality (MR) Assisted MitraClip Group: Patients undergoing MitraClip implantation with the assistance of MR technology, using Hololens 2.0 for three-dimensional visualization of DICOM images to enhance procedural precision and operator spatial awareness.
  Interventions: Procedure: MitraClip implantation
- Standard MitraClip Group: Patients undergoing MitraClip implantation using standard procedural methods without the assistance of MR technology.
  Interventions: Procedure: MitraClip implantation

INTERVENTIONS:
Procedure: MitraClip implantation — The MitraClip is used to catch the leaky parts of the mitral valve, and it is tested to ensure the leak is reduced.
  Other Names: TEER procedure

SUMMARY:
The study aims to evaluate the impact of mixed reality (MR) technology, particularly using Hololens 2.0 and specialized software for three-dimensional DICOM image visualization, on MitraClip implantation procedures. This preliminary case series includes a comparative analysis of four MitraClip implantations, assessing procedural efficiency, radiation exposure, and operator stress through both physiological and subjective measures.

DETAILED DESCRIPTION:
The advent of mixed reality (MR) technology, especially when integrated with Hololens 2.0 and specialized software for three-dimensional DICOM image visualization, offers promising avenues for enhancing precision and spatial awareness in interventional cardiology procedures. This case series aims to preliminarily evaluate the impact of MR on MitraClip implantation processes, setting the foundation for a comprehensive pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years
* Patients diagnosed with mitral valve regurgitation requiring MitraClip implantation
* Ability to provide informed consent and comply with study procedures

Exclusion Criteria:

* Patients with contraindications for MR technology (e.g., MRI incompatibility)
* Individuals unable to comply with study procedures due to physical or cognitive impairments
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult patients aged over 18 who require MitraClip implantation for the treatment of mitral valve regurgitation. These patients are selected from the patient pool at Hospital AGEL Trinec-Podlesi, Trinec, Czechia.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Operator stress indicator 1 | Measured pre-procedure, immediately post-procedure
  difference of cortisol levels in mmol/l
Operator stress indicator 2 | During the MitraClip implantation procedure, measured in real-time from the start to the completion of the procedure.
  heart rate variability of operator in BPM
Operator stress indicators 3 | During the MitraClip implantation procedure, measured in real-time from the start to the completion of the procedure.
  QTc interval in ms
Subjective assessments 1 | Administered immediately post-procedure.
  NASA TLX questionnaire with weighted score - method assesses work load on five 7-point scales
Subjective assessments 2 | Administered immediately post-procedure.
  STAI Y questionnaire with varies from a minimum score of 20 to a maximum score of 80
Subjective assessments 3 | Administered immediately post-procedure.
  SSQ questionnaire with assign a score from 0-3 for each of the sixteen items on the SSQ

SECONDARY OUTCOMES:
Procedural efficiency | From the beginning of the MitraClip implantation procedure until the completion of the procedure, measured in real-time, typically ranging from 1 to 3 hours.
  time of procedure
Radiation time exposure | From the start of the MitraClip implantation procedure until the end of fluoroscopy use, measured in real-time throughout the duration of the procedure, typically ranging from 30 to 120 minutes.
  Fluoroscopy Time (in minutes)
Radiation dose exposure | From the start of the MitraClip implantation procedure until the end of fluoroscopy use, measured in real-time throughout the duration of the procedure, typically ranging from 30 to 120 minutes.
  Dose Area Product (DAP) through the procedure in Gy·cm²

CONTACTS AND LOCATIONS:
Overall Officials: Otakar Jiravsky, MD, Study Director — Hospital Agel Trinec-Podlesi
Locations (1):
- Hospital AGEL Trinec-Podlesi a.s., Třinec, CZ, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The study plans to share de-identified individual participant data (IPD) to facilitate transparency and further research in the field of interventional cardiology and mixed reality (MR) technology applications. The shared data will be stripped of any personal identifiers to maintain participant confidentiality and adhere to data protection regulations.